CLINICAL TRIAL: NCT05247996
Title: TACE Combined With "Target Immune" Therapy for First-line Treatment Compared With Intravenous Chemotherapy in the Treatment of Unresectable Intrahepatic Cholangiocarcinoma: A Prospective, Multicenter, Open, Real-World Clinical Study
Brief Title: TACE Combined With "Target Immune" Therapy for First-line Treatment in the Treatment of Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZJLS-KLDMIR-22003
Record Dates: First submitted 2022-01-24; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-01

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Cholangiocarcinoma; Transcatheter arterial chemoembolization; Target therapy; Immune therapy; Systemic Intravenous Chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Immunotherapy, Active

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is an open-label study. The participants and investigators are not blinded, but the outcomes assessor are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcatheter arterial chemoembolization Combined With "Target Immune" Therapy (Experimental): Transcatheter arterial chemoembolization combined with immune checkpoint inhibitors and multi-target drugs was used for treatment.
  Interventions: Procedure: Transcatheter arterial chemoembolization; Drug: Multi-target Drug Therapy; Drug: Immunocheckpoint Inhibitor Therapy
- Traditional Systemic Intravenous Chemotherapy Group (Active Comparator): Traditional systemic intravenous chemotherapy with GEMOX regimen was used for comparison.
  Interventions: Procedure: Systemic Intravenous Chemotherapy

INTERVENTIONS:
Procedure: Transcatheter arterial chemoembolization — Treatment regimens have chosen "lipiodol-based" hepatic arterial chemoembolization, with lipiodol dosage varying from 5-20ml depending on tumor size. The chemotherapy drug is gemcitabine 1.0 combined with 100mg oxaliplatin, combined with 1/3 to 1 dose of solid embolic agent (the dosage is determined by the investigator based on the tumor size). After uniform emulsification, the drug is injected into the supplying blood vessels and stops when the intravascular blood flow is slow. Later, angiography is performed again, and the tumor staining disappears and the supplying artery is occlusions.
  CT or MRI scans are performed 4 to 6 weeks postoperatively to assess the presence of active lesions. Repeat TACE if active lesions are still present. The frequency of TACE treatment is determined by the investigator and is given according to the patient's condition, generally 2-4 times. The interval between TACE treatments is 30-45 days, with a maximum of six cycles.
  Other Names: TACE Thrapy
  Arms: Transcatheter arterial chemoembolization Combined With "Target Immune" Therapy
Drug: Multi-target Drug Therapy — Multi-target drugs (lenvatinib or donafenib) are selected at the patient's preference. Oral multitarget drugs are initiated 3-7 days after initial TACE treatment until tumor progression is assessed. The initial dose of lenvatinib is 8mg/ day (bodyweight < 60 kg) or 12 mg/ day (body weight≥60 kg); Donafenil 0.2g, twice a day, taken orally on an empty stomach. If the medication is missed, there is no need to take a refill and the next dose shall be taken at the usual time.
  Other Names: Target Therapy
  Arms: Transcatheter arterial chemoembolization Combined With "Target Immune" Therapy
Drug: Immunocheckpoint Inhibitor Therapy — Optional types of immune checkpoint inhibitors include Sintilimab injection and Tislelizumab injection. Treatment shall be based on the immune checkpoint inhibitors before enrollment, and it is not recommended to change the immune checkpoint inhibitors; Dosage: 200mg, iv, D1, every 21 days (Q3W), continuous until tumor progression.
  Other Names: Immune Therapy
  Arms: Transcatheter arterial chemoembolization Combined With "Target Immune" Therapy
Procedure: Systemic Intravenous Chemotherapy — GEMOX regimen (gemcitabine 1000mg/m2, oxaliplatin 100mg/m2) is given for systemic intravenous chemotherapy after the exclusion of contraindications for chemotherapy, and the presence of active lesions is assessed by laboratory and imaging examinations after every two courses of treatment. If active lesions remain, repeated systemic intravenous chemotherapy may be performed. The frequency of chemotherapy is determined by the investigator and is given according to the needs of the patient, usually 6 times with an interval of 21-28 days.
  Other Names: Traditional Chemotherapy
  Arms: Traditional Systemic Intravenous Chemotherapy Group

SUMMARY:
This study is a prospective, multicenter, open, real-world clinical study. All eligible patients were assigned to experimental group (TACE combined with multi-target drugs and PD-1 inhibitors), and control group (conventional intravenous chemotherapy), to explore the efficacy and safety of TACE combined with multi-target drugs and PD-1 inhibitors as first-line treatment compared with traditional systemic intravenous chemotherapy in the treatment of unresectable intrahepatic cholangiocarcinoma (ICC).

DETAILED DESCRIPTION:
This study is a prospective, multi-center, open, and double-arm clinical study in the real world, which belongs to a practical clinical trial. The type of comparison is the non-inferiority test. This study enrolls 98 patients with unresectable intrahepatic cholangiocarcinoma at multiple centers across the country. In the experimental group, 49 patients will receive TACE combined with immune checkpoint inhibitors and multi-target drugs; In the control group, 49 patients will receive traditional systemic intravenous chemotherapy with GEMOX regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients shall be older than 18 years old and have no gender limitation;
* Patients with intrahepatic cholangiocarcinoma confirmed by histopathology or clinical diagnosis and treatment standards who are inoperable or unwilling to undergo surgery at first diagnosis or who cannot be resected after recurrence;
* Patients with measurable lesions that can be observed and evaluated and whose diameter≥1cm are accurately measured by MRI enhancement or Computed Tomography (CT) enhancement according to mRECIST criteria;
* Patients with Child-Pugh A or B liver function grade and basically normal heart function;
* ECOG PS score≤1;
* Patients with expected survival > 3 months;
* Patients who have voluntarily participated in the study, signed informed consent, had good compliance, and cooperated with follow-up;
* There is no active HBV-DNA replication before enrollment (HBV-DNA<2000IU/mL), and HBV-positive patients have received anti-HBV treatment before enrollment.

Exclusion Criteria:

* Pregnant women, breast-feeding women or patients of childbearing age planning;
* Patients with severe heart, liver, and renal insufficiency and thyroid dysfunction;
* Patients scheduled for liver transplantation;
* Patients who have had or are currently suffering from other malignant tumors within five years, except cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumor;
* Patients with pleural effusion or ascites, causing respiratory syndrome (≥ CTCAE grade 2 dyspnea);
* Patients with unmitigated toxicity higher than CTCAE level 1 (5.0) due to any prior treatment;
* Patients with multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea, etc.);
* Patients with symptoms and signs of interstitial diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | The time from enrollment to tumor progression or death from any cause, whichever came first, measured in "months", assessed up to 2 years.
  The most common primary endpoint in cancer trials. The 6 months, 1 year, and 2 years progression-free survival

SECONDARY OUTCOMES:
Overall Survival | Time from randomization to death from any cause, in "months", assessed up to 2 years. For patients who are still alive at the time of data analysis, OS is calculated based on the date when the patient is last known to be alive.
  The best efficacy endpoint in cancer clinical trials.
Time To Tumor Untreatable Progression | The time interval between receiving TACE or intravenous chemotherapy and the patient's inability to receive further intra-arterial treatment, assessed up to 12 months.
  End point of antitumor drug trial.
Objective Response Rate | Proportion of patients who achieved complete remission (CR) or partial remission (PR) according to mRECIST criteria, assessed up to 12 months.
  Evaluation index of clinical efficacy of anticancer drugs.
Disease Control Rate | Proportion of patients with complete remission (CR), partial remission (PR), and stable disease (SD) according to mRECIST criteria, assessed up to 12 months.
  Evaluation index of clinical efficacy of anticancer drugs.
Duration of Overall Response | The time from the first assessment of the tumor as complete remission or partial remission to the first assessment as disease progression or death from any cause, assessed up to 12 months.
  Evaluation index of clinical efficacy of anticancer drugs.
The incidence of adverse events and serious adverse events | The time from randomization to every follow-up time, assessed up to 2 years.
  According to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xihui Ying, MD., Study Director — The Central Hospital of Lishui City

IPD SHARING:
Plan to Share IPD: Yes
Statistical analysis plan, informed consent form, and clinical study report can be shared with other researchers.
Supporting Information: SAP, ICF, CSR
Time Frame: Within six months after the trial is completed.
Access Criteria: Shared data is not available for downloading, but can only be browsed. To download the data, you must contact the researchers. Shared data does not provide any private information of the participants.

REFERENCES:
- [Background] Kelley RK, Bridgewater J, Gores GJ, Zhu AX. Systemic therapies for intrahepatic cholangiocarcinoma. J Hepatol. 2020 Feb;72(2):353-363. doi: 10.1016/j.jhep.2019.10.009. PMID 31954497
- [Background] Nathan H, Aloia TA, Vauthey JN, Abdalla EK, Zhu AX, Schulick RD, Choti MA, Pawlik TM. A proposed staging system for intrahepatic cholangiocarcinoma. Ann Surg Oncol. 2009 Jan;16(1):14-22. doi: 10.1245/s10434-008-0180-z. Epub 2008 Nov 6. PMID 18987916
- [Background] Zou L, Li X, Wu X, Cui J, Cui X, Song X, Ren T, Han X, Zhu Y, Li H, Wu W, Wang X, Gong W, Wang L, Li M, Lau WY, Liu Y. Modified FOLFIRINOX versus gemcitabine plus oxaliplatin as first-line chemotherapy for patients with locally advanced or metastatic cholangiocarcinoma: a retrospective comparative study. BMC Cancer. 2021 Jul 16;21(1):818. doi: 10.1186/s12885-021-08549-2. PMID 34266407
- [Background] Hu Y, Hao M, Chen Q, Chen Z, Lin H. Comparison of the efficacy and safety among apatinib plus drug-eluting bead transarterial chemoembolization (TACE), apatinib plus conventional TACE and apatinib alone in advanced intrahepatic cholangiocarcinoma. Am J Transl Res. 2020 Oct 15;12(10):6584-6598. eCollection 2020. PMID 33194055
- [Background] Wang L, Lin ZG, Ke Q, Lou JY, Zheng SG, Bi XY, Wang JM, Guo W, Li FY, Wang J, Zheng YM, Li JD, Cheng S, Zhou WP, Zeng YY. Adjuvant transarterial chemoembolization following radical resection for intrahepatic cholangiocarcinoma: A multi-center retrospective study. J Cancer. 2020 Apr 7;11(14):4115-4122. doi: 10.7150/jca.40358. eCollection 2020. PMID 32368294